CLINICAL TRIAL: NCT01435304
Title: The Effect of the Hemobag® Ultrafiltration System on Blood Conservation and Coagulation After Cardiopulmonary Bypass
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MaineHealth (Other)
Collaborators: Global Blood Resources, LLC (Other)
Responsible Party: Principal Investigator, Robert Kramer, MD, Director of Research and Quality Improvement Division of Cardiothoracic Surgery, MaineHealth
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB # 3914
Record Dates: First submitted 2011-09-09; First posted 2011-09-16 (Estimated); Results first posted 2018-05-02 (Actual); Last update posted 2018-06-06 (Actual); Status verified 2018-05

CONDITIONS: Blood Coagulation Disorders
MeSH Terms: conditions — Blood Coagulation Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hemobag® (Experimental): Hemobag® method of returning residual CPB blood (study group)
  Interventions: Device: method of returning residual CPB blood ( Hemobag®)
- cell saver (No Intervention): Standard method of returning the residual pump volume to the patient as washed, centrifuged cells (control group)

INTERVENTIONS:
Device: method of returning residual CPB blood ( Hemobag®) — The Hemobag® is a collection reservoir used to facilitate ultrafiltration of the CPB circuit after the patient has been disconnected from CPB).
  Other Names: Hemobag®
  Arms: Hemobag®

SUMMARY:
This proposal is designed to mitigate hemodilution (blood diluted with an electrolyte solution) and loss of plasma proteins responsible for normal blood clotting as well as platelets at the completion of cardiopulmonary bypass (CPB). The Hemobag® system is a device qualified by the US Food and Drug Administration (FDA). Many cardiac centers, such as Englewood Hospital and Medical Center in Englewood NJ are using the Hemobag® system for Jehovah's witnesses and other patients who go to that center for bloodless cardiac surgery (cardiac surgery performed without the use of blood or blood products). The system is designed to filter excessive water from blood left in the heart lung machine (cardiopulmonary bypass) after it is separated from the patient during the performance of cardiac surgery. Consequently the likelihood of excessive post-operative bleeding and transfusion with allogeneic blood (blood bank blood from donors) is decreased.

DETAILED DESCRIPTION:
Background:

Cardiopulmonary bypass (CPB) consists of an extracorporeal (outside of the body) circuit which allows the circulation and oxygenation of blood during cardiac surgery. The circuit includes an oxygenator, a reservoir and tubing, all of which needs to be primed with a balanced electrolyte solution. Prior to initiating CPB, the venous and arterial ends of the CPB circuit are appropriately attached to the patient. The volume of the circuit is usually 1.5 liters which is equivalent to 30-38% of a typical patient's total blood volume that is generally between 4 and 5 liters.

When CPB is initiated, the patient's blood is mixed and diluted by the CPB priming fluid. Consequently, when the operation is completed and the CPB is discontinued, the content of the CPB circuit consists of the patient's diluted whole blood. The standard practice is to return as much of this hemodiluted CPB contents as the patient will accommodate and process the rest of the contents of the circuit with a cell washer and return packed red blood cells to the patient.

When the cell washer is used, plasma proteins, clotting factors and platelets are not returned to the patient. An alternate approach would be to use an ultrafiltration device to remove this non-cellular water and preserve proteins,

clotting factors and platelets as well as red blood cells that can then be returned to the patient. This alternate approach is the basic principle of the Hemobag®, an ultrafiltration technology and method.

Ultrafiltration is a well documented technique usually used in-line (interposed in the circuit) during CPB. The Hemobag® is a collection reservoir used to facilitate ultrafiltration of the CPB circuit after the patient has been disconnected from CPB). It represents a novel and safe modification of the modified ultrafiltration system (MUF). MUF is a technique commonly used in cardiac surgery for many years, especially with smaller hemodiluted patients, and mainly in the pediatric population.

The focus of the Hemobag® system is on whole blood volume recovery as opposed to red cell volume recovery only, and helping to satisfy the requirements of the patient after CPB has been discontinued: hemostasis, reversal of dilutional effects, and returning back to homeostasis, which is the normal physiologic and metabolic status of the patient.

The investigators hypothesize that the Hemobag® method of returning residual CPB blood is superior to the current practice of cell washing and concentration. This hypothesis is based on previous studies that have shown that the ultrafiltrated whole blood product is superior to the cell-washed RBC product. The main purpose of this study is to discover the differences in outcome measures when, at the end of CPB, the residual diluted pump blood is processed by either cell washing or by the Hemobag® method. The null hypothesis states that there would be no difference in post-operative patient outcomes when residual pump blood is processed by either a cell washing method or the Hemobag® protocol.

Pilot Study:

The investigators did an Maine Medical Center (MMC) Institutional Review Board (IRB)-approved pilot study in March 2011 which consisted of ten (10) cases in order to confirm the significant treatment effect shown in other studies and to familiarize the team with the Hemobag® system. Outcome metrics included chest catheter drainage in the first 24 hours post-operative, allogeneic blood component requirements (red blood cells (RBC's), platelets, plasma), platelet counts, evidence of acute kidney injury by the Acute Kidney Injury Network (AKIN) definition, mortality, stroke, and requirements for inotropic support on the second post-operative day. The results of the pilot study showed a promising trend with regard to less chest catheter drainage and higher platelet counts.

Materials and Methods and Analysis:

The investigators propose to do a randomized, controlled trial comparing the two methods as described above: The standard method of returning the residual pump volume to the patient as washed, centrifuged cells (control group) and the Hemobag® method of returning residual CPB blood (study group).

Outcome metrics will be the same as they were for the pilot study:

(1) Chest catheter drainage in the first 24 hours post-operative; (2) Allogeneic blood component requirements (RBC's, platelets, plasma); (3) Pre and post operative platelet counts; (4) Evidence of acute kidney injury by AKIN definition; (5) Mortality; (6) Stroke; (7) Requirements for inotropic support on the 2nd post-operative day.

The investigators propose to enroll 100 patients, 50 in the control group and 50 in the study group. The study will be limited to adults (18 years and older) who have heart surgery (valve and /or coronary) using CPB who do not have anemia or coagulation disorders preoperatively.

An interim analysis will be performed by an independent, unblended analyst to determine efficacy and safety half way through the study (50 patients). Terminating the study early would be a consideration if one group were clearly superior to the other or if there were safety issues. In the event that there are no concerns regarding superiority or safety, the study would continue until the entire sample size has been studied. The results of the interim analysis will be submitted to the IRB.

Conclusion:

There are a number of intra-operative blood management strategies in cardiac surgery and the salvage of post-CPB whole blood using ultrafiltration from the CPB circuit is emerging as one of the most significant contributors to reducing allogeneic blood component use in cardiovascular surgery. The investigators hypothesize that the Hemobag® method of returning residual CPB blood is superior to the current practice of cell washing and concentration and more expeditious than modified ultrafiltration (MUF).

ELIGIBILITY:
Inclusion Criteria:

All adult cardiac surgery patients (age 18 or older) Cardiopulmonary bypass

Exclusion Criteria:

Patients under age 18 Off pump surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-09; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Kramer, MD, Principal Investigator — MaineHealth
Locations (1):
- Maine Medical Center, Portland, Maine, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Hemobag® | Cell Saver
Started | 50 | 50
Completed | 50 | 50
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Hemobag® | Cell Saver | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.4 (10.5) | 63.3 (15.3) | 63.8 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 7 | 22
  Male | 35 | 43 | 78
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 50 | 50 | 100

OUTCOME MEASURES:

1. Primary Outcome: Amount of Chest Catheter Drainage 24 Hours Postoperatively
Description: Chest catheters are placed in the mediastinum and sometimes pleural space(s) to collect shed mediastinal blood in the first 24 hours post operative cardiac surgery
Time Frame: Total amount for the first 24 hours postoperative
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Hemobag® | Cell Saver
Number analyzed (Participants) | 50 | 50
mL | 766 (845) | 626 (427)

2. Secondary Outcome: Number of Participants Which Had Blood Products Transfused (RBC's, Platelets, FFP)
Description: These blood components can be a metric of the success of achieving a satisfactory coagulation status.
Time Frame: All blood products transfused during index admission, an expected average of 7 days, with the exception of preoperative transfusions.
Measure: Count of Participants; unit: Participants
Arm/Group | Hemobag® | Cell Saver
Number analyzed (Participants) | 50 | 50
Participants | 8 | 6

3. Secondary Outcome: Number of Participants With Acute Kidney Injury (AKI)
Description: Using the Acute Kidney Injury Network (AKIN) definition of a 0.03mg/dL increase in serum creatinine within 48 hours of surgery, serial postoperative creatinines will reflect the presence of AKI when compared with the baseline creatinine.
Time Frame: All creatinines will be recorded and assessed during the entire index admission in order to compare postoperative to preoperative baseline creatinine, an expected average of 7 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Hemobag® | Cell Saver
Number analyzed (Participants) | 50 | 50
Participants | 6 | 6

4. Secondary Outcome: Number of Participants With a Mortality
Description: Patients will be followed until hospital discharge
Time Frame: Index admission postoperative until the time of discharge, an expected average of 7 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Hemobag® | Cell Saver
Number analyzed (Participants) | 50 | 50
Participants | 2 | 1

5. Secondary Outcome: Number of Participants With Stroke
Description: Any neurological defect according to Society of Thoracic Surgery (STS) definition
Time Frame: Index admission postoperative until the time of discharge, an expected average of 7 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Hemobag® | Cell Saver
Number analyzed (Participants) | 50 | 50
Participants | 0 | 2

6. Secondary Outcome: Number of Participants on Vasoactive Drugs at 48 Hours Post op Point
Description: This metric is a surrogate for low output failure and /or vasoplegia depending upon whether inotropes or vasoconstrictors are used.
Time Frame: Any intravenous vasoactive drug being used at the 48 hour time point postoperative
Measure: Count of Participants; unit: Participants
Arm/Group | Hemobag® | Cell Saver
Number analyzed (Participants) | 50 | 50
Participants | 12 | 14

ADVERSE EVENTS:
Arm/Group | Hemobag® | Cell Saver
All-Cause Mortality (participants affected / at risk) | 2/50 | 1/50
Serious Adverse Events (participants affected / at risk) | 0/50 | 2/50
Other Adverse Events (participants affected / at risk) | 12/50 | 14/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hemobag® (N=50) | Cell Saver (N=50)
Stroke (Nervous system disorders) | 0 (0) | 2 (2) — Any neurological defect according to Society of Thoracic Surgery (STS)...
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hemobag® (N=50) | Cell Saver (N=50)
Low output failure (Cardiac disorders) | 12 (12) | 14 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No